CLINICAL TRIAL: NCT05167227
Title: The Long COVID and Fatiguing Illness Recovery Program - A Pragmatic, Quality Improvement, Professional Cluster, Randomized Controlled Trial.
Brief Title: Does a Technology Enabled Multi-disciplinary Team-based Care Model for the Management of Long COVID and Other Fatiguing Illnesses Improve Clinical Care of Patients and Represent a Sustainable Approach Within a Federally Qualified Health Center?
Acronym: LC&FIRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Family Health Centers of San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2021-0241
Record Dates: First submitted 2021-12-17; First posted 2021-12-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; Post-acute Sequelae of SARS-COV-2 Infection; Post COVID-19 Condition
Keywords: Long COVID; ME; CFS; PASC; PCC
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: 20 consenting clinicians across primary care clinics at FHCSD will be randomized at a ratio of 1:1 to either participate in 1) weekly teleECHO sessions with monthly interactive webinars and quarterly short courses or 2) monthly interactive webinars and quarterly short courses alone (a control group). Throughout participation, the investigators expect that the clinicians will provide care for approximately 856 FHCSD patients diagnosed with PASC, ME/CFS, or OPIFI (approximately 42 patients per clinician). The clinicians will be consented and will receive exposure to intervention components (i.e., a professional cluster). Therefore, patient outcomes derived from routine clinical care will be evaluated according to the study arm of their respective clinicians.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation will be concealed from all investigators and staff until the study group is assigned. Only the study manager and research assistants involved in the delivery of the intervention components will subsequently be made aware of allocation. It is not possible to mask participating clinicians, however, patients of participating clinicians will not have knowledge of their clinicians potential participation in weekly teleECHO sessions, monthly interactive webinars, and quarterly short courses. All staff that are involved in the collection of data and investigators that conduct analyses will remain blinded to allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The Control arm participates in monthly interactive webinars and quarterly short courses.
  Monthly interactive webinars will offer brief didactic presentations by SMEs, examples of models of care, and a facilitated Q&A. These webinars will be convened to rapidly disseminate findings and emerging best practices to a large-scale, national audience.
  Quarterly short courses will be developed to summarize key findings from past weekly teleECHO sessions. These quarterly short courses will be formatted as a learning module with the use of presentation slides and videos online that are accessible asynchronously.
- Intervention (Experimental): The Intervention arm participates in weekly teleECHO sessions with monthly interactive webinars and quarterly short courses.
  Interventions: Other: Extension for Community Healthcare Outcomes

INTERVENTIONS:
Other: Extension for Community Healthcare Outcomes — ECHO is a technology enabled multi-disciplinary team-based care model centered on case-consultation and peer-to-peer sharing of emerging best practices (i.e., teleECHO) to support management of complex cases associated with Long COVID, ME/CFS, and other PIFI.
  Other Names: ECHO
  Arms: Intervention

SUMMARY:
The primary objective of the present research is to determine the effectiveness of Family Health Center of San Diego's Long COVID and Fatiguing Illness Recovery Program (LC&FIRP) on clinician- and patient-level outcomes. LC&FIRP is comprised of a teleECHO program focused on multi-specialty case-consultation and peer-to-peer sharing of emerging best practices to support management of complex cases associated with Long COVID, Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS), and other post-infectious fatiguing illnesses (PIFI). Our secondary objective is to determine the feasibility, acceptability, and sustainability of LC&FIRP. Our findings should provide a fuller understanding of the potential impact of innovative technology enabled multi-disciplinary team-based care models in low-resource, community-based primary care settings.

DETAILED DESCRIPTION:
The primary objective of the present research is to determine the effectiveness of FHCSD's Long COVID and Fatiguing Illness Recovery Program (LC&FIRP) on clinician- and patient-level outcomes. LC&FIRP is comprised of a teleECHO program focused on multi-specialty case-consultation and peer-to-peer sharing of emerging best practices to support management of complex cases associated with Long COVID, ME/CFS, and other PIFI. Our secondary objective is to determine the feasibility, acceptability, and sustainability of LC&FIRP. Our findings should provide a fuller understanding of the potential impact of innovative technology enabled multi-disciplinary team-based care models in low-resource, community-based primary care settings. This study will provide much needed high-quality evidence on the effectiveness of a technology enabled multi-disciplinary team-based care model for the management of Long COVID, ME/CFS, and other PIFI within a community clinic setting, while simultaneously providing evidence regarding the feasibility, acceptability, and sustainability of the approach. Given that LC&FIRP includes a teleECHO program that is case-based, interactive, and occurs in real-time, it has a set of distinct advantages to the traditional practice of sequential in-person specialty referrals to address complex patient cases. The investigators hypothesize that clinician exposure to weekly teleECHO sessions with monthly interactive webinars and quarterly short courses will significantly improve clinician- and patient-level outcomes compared to clinician exposure to monthly interactive webinars and quarterly short courses alone.

The investigators will evaluate LC&FIRP using an effectiveness-implementation hybrid type 2 design. Specifically, the investigators will conduct a two-arm, single-blind, pragmatic, quality improvement, professional cluster, randomized controlled trial. The target for weekly teleECHO sessions, monthly interactive webinars, and quarterly short courses are licensed health care professionals. Therefore, the present research will include professional clusters that will consist of primary care physicians, physician assistants, and nurse practitioners at FHCSD caring for patients who have had persistent symptoms and a decline in health-related quality of life associated with Long COVID, ME/CFS, and/or other PIFI.

20 consenting clinicians across primary care clinics at FHCSD will be randomized at a ratio of 1:1 to either participate in 1) weekly teleECHO sessions with monthly interactive webinars and quarterly short courses or 2) monthly interactive webinars and quarterly short courses alone (a control group). All clinicians will have the option to receive continuing medical education credit for the educational sessions they engage in. Throughout participation, the investigators expect that the clinicians will provide care for approximately 856 FHCSD patients diagnosed with Long COVID, ME/CFS, or other PIFI (approximately 42 patients per clinician). The clinicians will be consented and will receive exposure to intervention components (i.e., a professional cluster). Therefore, patient outcomes derived from routine clinical care will be evaluated according to the study arm of their respective clinicians. Outcomes will be measured at 3-, 6-, 9-,12-, 18-, 24-, and 30-months post-baseline for clinicians and for patients at 3-, 6-, 9-, and 12-months post assignment to a participating clinician.

Inclusion criteria for clinicians includes 1) being employed by FHCSD for clinical care delivery, 2) being a licensed primary care physician, physician assistant, or nurse practitioner, 3) caring for patients who have had persistent symptoms and a decline in health-related quality of life associated with Long COVID, ME/CFS, and/or other PIFI, and 4) being willing and able to actively participate in LC&FIRP. There are no exclusion criteria. FHCSD medical leadership has verbally extended an invitation to the approximately 200 eligible clinicians at FHCSD to participate in LC&FIRP (a follow-up email will also be sent). Those who are interested will provide written informed consent, complete a baseline survey, and will be randomized to one of the two study arms. An electronic randomization list will be generated using the latest version of the statistical software platform R (version 3.3.2, http://www.r-project.org). The list will be securely integrated into the cloud-based Research Electronic Data Capture (REDCap) tool. Allocation will be concealed from all investigators and staff until the study group is assigned. Only the study manager and research assistants involved in the delivery of the intervention components will subsequently be made aware of allocation. It is not possible to mask participating clinicians, however, patients of participating clinicians will not have knowledge of their clinicians potential participation in weekly teleECHO sessions, monthly interactive webinars, and quarterly short courses. All staff that are involved in the collection of data and investigators that conduct analyses will remain blinded to allocation throughout the study.

Clinician participation in this study is voluntary. Participating clinicians may decide not to participate or may leave the study at any time. This decision will not result in any penalty or loss of benefits to which they are entitled. Information that has already been collected may still be used, but no new information will be collected. The withdrawal reason and the withdrawal date will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for clinicians includes 1) being employed by FHCSD for clinical care delivery, 2) being a licensed primary care physician, physician assistant, or nurse practitioner, 3) caring for patients who have had persistent symptoms and a decline in health-related quality of life associated with PASC, ME/CFS, and/or OPIFI, and 4) being willing and able to actively participate in LC&FIRP.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | During 12 months of follow-up
  Patient baseline and quarterly surveys

SECONDARY OUTCOMES:
Patient symptom checklist with associated severity for those present | During 12 months of follow-up
  Patient baseline and quarterly surveys, None, Mild, Moderate, Severe
If symptom is present, has patient experienced this in the past month | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes/No
If symptom is present, how long has patient experienced this symptom | During 12 months of follow-up
  Patient baseline and quarterly surveys, Under 3 Months, 3 Months or longer
If symptom is present, did patient have this symptom before the patient tested positive for COVID-19? | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes/No
If symptom is present, during the past month how often have the patient had this symptom? | During 12 months of follow-up
  Patient baseline and quarterly surveys with use of Likert scale
If symptom is present during the past month, how bad was this symptom? | During 12 months of follow-up
  Patient baseline and quarterly surveys with use of Likert scale
For symptoms present, do any of them get worse for at least 24 hours after engaging in activities (physical or mental) that patient was used to doing with no problems? | During 12 months of follow-up
  Patient baseline and quarterly surveys with Yes/No/Not Applicable/Don't Know
If fatigue, tiredness, or exhaustion is present, doesn't patient describe it as feeling it come on all of a sudden, or slowly over time | During 12 months of follow-up
  Patient baseline and quarterly surveys with All of sudden, Slowly over time, Not applicable, Don't know
If fatigue present, what month and year did the fatiguing illness begin? | During 12 months of follow-up
  Patient baseline and quarterly surveys, estimated month and year
When fatigued, does rest make patient's fatigue better? | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes a lot, Yes a little, No not very much, Not applicable, Don't know
When fatigued, has this fatigue substantially limited the patient's ability to occupational, educational, social, or personal activities? | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes, No, Not applicable, Don't know
Patient's medical history check-list | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes, No, Unsure
Patient's dietary restrictions | Through study referral period, an average of 12 weeks
  Patient baseline survey, No, Vegan, Vegetarian, Ketogenic, Gluten-free, Dairy-free, Intermittent fasting, Other
Patient's food allergies or other food intolerances | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes/No
Has patient's employment been impacted due to contracting COVID-19? | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes, No
Patient's frequency to complete 150-minutes per week of moderate-intensity physical activity (like a brisk walk, slow biking, gardening, or ballroom dancing) prior to contracting COVID-19 | Through study referral period, an average of 12 weeks
  Patient baseline survey, Every week, Most weeks, Some weeks, Very few weeks, Never, I do not know
Patient's frequency to complete 150-minutes per week of vigorous-intensity physical activity (like running, swimming laps, competitive sports, or fast bicycling) prior to contracting COVID-19 | Through study referral period, an average of 12 weeks
  Patient baseline survey, Every week, Most weeks, Some weeks, Very few weeks, Never, I do not know
Did patient receive a COVID-19 PCR (nasal swab) test | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes/No
Did patient receive a COVID-19 antibody test | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes/No
Patient symptom onset | Through study referral period, an average of 12 weeks
  Patient baseline survey, Date
Patient reported medications used for COVID-19 symptoms | Through study referral period, an average of 12 weeks
  Patient baseline survey, free text
Patient reported prescribed supplementary oxygen support | Through study referral period, an average of 12 weeks
  Patient baseline survey, Yes/No
Patient reported admittance to hospital due to COVID-19 | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes/No
Do any of the following activities exacerbate patients symptoms: Physical exertion, Diet Changes, Big Meal, Dehydration, Weather changes (hot and humid), Tight clothing, Stress or anxiety, Pre Menstrual period, Menstrual period, Alcohol consumption | During 12 months of follow-up
  Patient baseline and quarterly surveys, Yes/No
Does patient feel fully recovered from COVID-19 | During 9 months of follow-up
  Patient quarterly surveys, Yes/No
Currently minutes per week of moderate-intensity physical activity patient does (like a brisk walk, slow biking, gardening, or ballroom dancing) | During 9 months of follow-up
  Patient quarterly surveys, free text
Currently minutes per week of vigorous-intensity physical activity patient does (like running, swimming laps, competitive sports, or fast bicycling) | During 9 months of follow-up
  Patient quarterly surveys, free text
Patient Health Questionnaire (PHQ)-2 | During 12 months of follow-up
  Patient baseline and quarterly surveys
Patient Health Questionnaire (PHQ)-9 (if applicable) | During 12 months of follow-up
  Patient baseline and quarterly surveys
PROMIS Dyspnea Functional Limitations and Severity Short Forms | During 12 months of follow-up
  Patient baseline and quarterly surveys
PROMIS Applied Cognition Abilities and General Concerns Short Forms | During 12 months of follow-up
  Patient baseline and quarterly surveys
Generalized Anxiety Disorder (GAD)-7 | During 12 months of follow-up
  Patient baseline and quarterly surveys
2-minute step test | During 12 months of follow-up
  Physical Therapy assessment with patient
30 sec sit to stand test | During 12 months of follow-up
  Physical Therapy assessment with patient
Grip strength | During 12 months of follow-up
  Physical Therapy assessment with patient
Functional Gait Assessment | During 12 months of follow-up
  Physical Therapy assessment with patient
Balance tasks | During 12 months of follow-up
  Physical Therapy assessment with patient
Post-exertional malaise follow-up | Per Physical Therapy encounter after PT assessment
  Follow-up Physical Therapy appointment with patient, Not at all, A little bit, Somewhat, Quite a bit, Very much

OTHER OUTCOMES:
Knowledge improvement of appropriate PASC diagnosis as a result of participation in randomized arm (teleECHO or monthly webinar) | During 37 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Knowledge improvement of effective PASC care and treatment as a result of participation in randomized arm (teleECHO or monthly webinar) | During 37 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Knowledge improvement of approaches for complex cases of PASC as a result of participation in randomized arm (teleECHO or monthly webinar) | During 37 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities related to identify tools and methods for PASC care | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to diagnose patients with PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to screen for co-morbidities of PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to generate a patient-specific treatment plan for patients with PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities related to to implement a patient-specific treatment plan for patients with PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to select appropriate special or diagnostic tests for PASC patients | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to interpret special or diagnostic test results for my PASC patients | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to provide appropriate patient education about their PASC condition | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to educate clinic staff about PASC care | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to address PASC patients using a multidisciplinary approach | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to assess and manage concerns that PASC patients face | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to assess severity of disease in patients with PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Self-efficacy in abilities to deal with complex cases of PASC | During 37 months of follow-up
  Clinician baseline and quarterly follow-up survey with use of Likert scale agreement
Utility of an encountered case presented during randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey Yes/No
Overall satisfaction with randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Satisfaction to recommend to colleague randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale likelihood
Satisfaction to participate in future randomized arm (teleECHO or monthly webinar) again | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale likelihood
Changes to practice in helping colleague with information learned from randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey Yes/No
Changes to practice by participating in randomized arm (teleECHO or monthly webinar) to understand further monitoring and follow-up plan | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Changes to practice by participating in randomized arm (teleECHO or monthly webinar) to develop more appropriate treatment plans | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Changes to practice by participating in randomized arm (teleECHO or monthly webinar) to have a better understanding of underlying disease process and the role of specialist referral | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Changes to practice by participating in randomized arm (teleECHO or monthly webinar) to more independently manage my PASC patients without referral to a specialist | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement
Changes to practice by participating in randomized arm (teleECHO or monthly webinar) to apply specialist recommendations to patient care. | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement and free text
Unable to apply learnings from randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey with use of Likert scale agreement and free text
Other changes to practice by participating in randomized arm (teleECHO or monthly webinar) | During 34 months of follow-up
  Clinician quarterly follow-up survey with free text
Knowledge gained about topic presented during teleECHO before and after | During 37 months after each weekly ECHO session
  Clinician intervention teleECHO survey
Knowledge gained about topic presented during teleECHO before and after | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale knowledge
Satisfaction with stated objectives being met | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Satisfaction with session delivering balanced and objective, evidence-based content | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Satisfaction with pace of session | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Satisfaction with opportunities to ask questions | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Satisfaction with organization of the presenters' presentations | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Satisfaction with presenters' ability to clearly communicate | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale quality
Desired content for future sessions | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey, free text
Satisfaction with source evidence presented | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey Yes/No
Satisfaction with commercial bias present | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey Yes/No and free text
Recommendations for program improvement | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey free text
Relevance of session to clinicians current work | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale relevance
Intent to change practice based on learnings from session | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey Yes/No and free text
Best part of session | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey free text
Worst part of session | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey free text
Recommend this session to a colleague | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey with use of Likert scale likelihood
Changes to practice planned | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey free text
If no changes to practice are planned, barriers | Through study completion, an average of 37 months
  Clinician intervention teleECHO survey free text
Participating clinician retention | Semi-annually during 37 months of follow-up
  Mean number of months clinicians participate in the trial (intervention and control groups)
Participating clinic settings | Semi-annually during 37 months of follow-up
  Number of clinic settings in which providers see patients (intervention and control groups)
Participation in intervention | Weekly during 37 months of follow-up
  Number of weekly sessions each RCT (intervention) provider attends, and mean number
Exposure of weekly teleECHO topics | Weekly during 37 months of follow-up
  Number of topics covered in Weekly ECHO sessions RCT (intervention) provider attends
Monthly webinar attendance | Monthly during 37 months of follow-up
  Number of monthly webinars RCT providers attends
Quarterly short course attendance | Quarterly during 37 months of follow-up
  Number of quarterly short courses RCT providers attends
Exposure of monthly webinar topics | Monthly during 37 months of follow-up
  Number of topics covered in monthly webinars provider attends
Exposure of quarterly short course topics | Quarterly during 37 months of follow-up
  Number of topics covered in quarterly short courses provider attends
Participation in case consultation | Quarterly during 37 months of follow-up
  Number of patient cases presented by RCT (intervention) provider
Participation in post-session survey | Weekly during 37 months of follow-up
  Proportion of participants that complete each session poll (disaggregated by monthly webinar, weekly session, RCT vs. non-RCT provider)
Volume of total patient case load | Monthly during 37 months of follow-up
  Number of patients seen by RCT provider, and mean number (intervention and control)
Volume of PASC patient case load | Monthly during 37 months of follow-up
  Number of PASC patients seen by RCT provider, and mean number (intervention and control)
Volume of patient referrals to specialists | Monthly during 37 months of follow-up
  Number of referrals to specialists by RCT provider, and mean number (intervention and control)
Application of specialist recommendations | Quarterly during 37 months of follow-up
  Number of specialist recommendations applied by RCT (intervention) providers from weekly ECHO sessions
Average consultation duration | Monthly during 37 months of follow-up
  Mean duration of consultation for PASC patients by RCT providers, intervention and control
Volume of specialists seen by patients | Monthly during 37 months of follow-up
  Number of specialists seen by patient
Specialty types patient was exposed to | Monthly during 37 months of follow-up
  Number of specialty types the patient was exposed to
Clinician session drop-off | Weekly during 37 months of follow-up
  How long an (intervention) provider attended an ECHO session
Quarterly attendance | Quarterly during 37 months of follow-up
  Number of individuals who attended and watched short course
Clinician satisfaction with series | Up to 8 weeks after end of study
  Interview with Likert satisfaction
Clinician overall best part of series | Up to 8 weeks after end of study
  Interview
Clinician overall worst part of series | Up to 8 weeks after end of study
  Interview
Clinician challenges in participating | Up to 8 weeks after end of study
  Interview
Perceived change in the relationship between clinicians and specialists in panel as a result of this series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Clinician barriers to sustained participation in series | Up to 8 weeks after end of study
  Interview
Did clinician experience an improvement in the number of PASC patients they could manage at any given time as a result of the series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinicians experience an increase in PASC patients in their panel composition over time as a result of participation in the series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinic directors observe an increase in PASC patients in the clinicians panel composition over time as a result of their participation in the series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinicians experience an improvement in the quality of care for patients as a result of participating in the series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinic directors observe an improvement in the quality of care for patients as a result of a clinician participating in the series? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinicians participating influence other providers in their clinic? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Did clinic directors observe clinicians who participated in the series influence other providers within the clinic? | Up to 8 weeks after end of study
  Interview, Yes/No with free response
Clinician benefits gained from participating in the series | Up to 8 weeks after end of study
  Interview, free response
Clinician recommendations for improving the scalability or sustainability of this model | Up to 8 weeks after end of study
  Interview, free response
Clinic directors recommendations for improving the scalability or sustainability of this model | Up to 8 weeks after end of study
  Interview, free response

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ramers, MD, Principal Investigator — Family Health Centers of San Diego; Job Godino, PhD, Principal Investigator — Family Health Centers of San Diego
Locations (1):
- Family Health Centers of San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godino JG, Samaniego JC, Sharp SP, Taren D, Zuber A, Armistad AJ, Dezan AM, Leyba AJ, Friedly JL, Bunnell AE, Matthews E, Miller MJ, Unger ER, Bertolli J, Hinckley A, Lin JS, Scott JD, Struminger BB, Ramers C. A technology-enabled multi-disciplinary team-based care model for the management of Long COVID and other fatiguing illnesses within a federally qualified health center: protocol for a two-arm, single-blind, pragmatic, quality improvement professional cluster randomized controlled trial. Trials. 2023 Aug 12;24(1):524. doi: 10.1186/s13063-023-07550-3. PMID 37573421